CLINICAL TRIAL: NCT03199911
Title: The Role of Topical Antibiotic Prophylaxis in Eyelid Surgery
Brief Title: Topical Antibiotic Prophylaxis for Eyelids
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 17-22309
Record Dates: First submitted 2017-06-08; First posted 2017-06-27 (Actual); Results first posted 2020-07-21 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Antibiotic Side Effect; Eyelid; Wound; Eyelid Diseases; Surgical Wound Infection; Surgical Wound, Recent; Surgical Incision; Skin Cancer Face; Antibiotic Allergy; Surgical Site Infection
MeSH Terms: conditions — Wounds and Injuries; Eyelid Diseases; Surgical Wound Infection; Surgical Wound | interventions — Erythromycin; Bacitracin

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to one of two intervention arms (i.e. antibiotic ointment vs. placebo artificial tear ointment) and will not at any point cross over to the other arm.
Masking Description: Randomization to one of two intervention arms (i.e. antibiotic ointment vs. placebo artificial tear ointment) will be performed prior to study recruitment by REDCap software. Patients' randomization assignments will be revealed at the initial pre-operative visit or at time that procedure consent is obtained; the study team will not be aware of a subject's randomization assignment prior to that time.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Topical Antibiotic Ointment (Experimental): Intervention: 200 patients in the antibiotic arm will receive either erythromycin or bacitracin, based on allergies, surgeon preference, and antibiotic availability. If neither antibiotic is obtainable by the patient, bacitracin polymyxin will be prescribed instead. Antibiotic ointment is to be applied to the surgical incision(s) 4 times daily for 1 week.
  Interventions: Drug: Topical Antibiotic Product
- Topical Non-Antibiotic Ointment (Placebo Comparator): Intervention: 200 patients in the placebo group will receive mineral oil/petrolatum-based artificial tear ointment to be applied to the surgical incision(s) 4 times daily for 1 week.
  Interventions: Drug: Topical Non-Antibiotic Ointment

INTERVENTIONS:
Drug: Topical Antibiotic Product — Topical antibiotic ointment will be erythromycin or bacitracin. If the patient cannot obtain either (e.g. lack of availability at the pharmacy), bacitracin polymyxin will be prescribed. Allergy to all 3 study drugs means that a patient will be excluded from the study.
  Other Names: Erythromycin, Bacitracin, Polysporin-Bacitracin
  Arms: Topical Antibiotic Ointment
Drug: Topical Non-Antibiotic Ointment — Mineral oil/petrolatum-based artificial tear ointment.
  Other Names: Refresh PM
  Arms: Topical Non-Antibiotic Ointment

SUMMARY:
The investigators propose a prospective randomized control trial testing the hypothesis that routine topical antibiotic prophylaxis does not significantly reduce the rate of infection after eyelid surgery.

DETAILED DESCRIPTION:
The use of prophylactic topical antibiotic therapy after eyelid surgery is widespread. Due to increasing antibiotic resistance, antibiotic-related complications, and healthcare costs, the investigators wish to determine whether prophylactic post-operative antibiotic ointment is truly necessary. After all, existing dermatology literature currently recommends against the routine use of antibiotic ointment after various surgical procedures (e.g. Mohs surgery). The investigators aim to perform a prospective randomized control trial at the University of California, San Francisco. The investigators aim to recruit a total of 400 oculoplastics patients undergoing eyelid surgery or surgery involving peri-orbital incisions from 2017 through 2019.

ELIGIBILITY:
Inclusion Criteria:

Patients aged 18 and older who are undergoing various eyelid procedures in an office, ambulatory care center, or operating room including but not limited to:

* blepharoplasty (upper and lower lids);
* ectropion repair;
* entropion repair;
* external dacryocystorhinostomy;
* external levator resection;
* eyelid lesion removal and/or biopsy;
* eyelid reconstruction and defect repair including after Mohs surgery;
* fat pad excision (upper and lower lids);
* gold or platinum weight implantation;
* internal levator resection;
* lateral tarsal strip;
* orbital fracture repair requiring periorbital incisions;
* orbitotomy requiring periorbital incisions;
* tarsorrhaphy;
* wedge excision.
* Patients undergoing repeat procedures will also be included.

Exclusion Criteria:

* Patients aged younger than 18 years old who are undergoing the above eyelid procedures in an office, ambulatory care centers, operating rooms;
* patients undergoing chalazion removal;
* patients who have had previous wound infections at the site of the procedure;
* patients with oral or IV antibiotic use within 10 days prior to procedure;
* patients requiring IV antibiotics during the procedure;
* patients with grossly contaminated or inflamed wounds;
* patients with human or animal bites, patients with wounds resulting from trauma
* patients allergic to all study drug options.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 401 (Actual)
Dates: Start 2017-10-02 (Actual); Primary Completion 2019-11-14 (Actual); Study Completion 2019-11-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Kersten, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fay A, Nallasamy N, Bernardini F, Wladis EJ, Durand ML, Devoto MH, Meyer D, Hartstein M, Honavar S, Osaki MH, Osaki TH, Santiago YM, Sales-Sanz M, Vadala G, Verity D. Multinational Comparison of Prophylactic Antibiotic Use for Eyelid Surgery. JAMA Ophthalmol. 2015 Jul;133(7):778-84. doi: 10.1001/jamaophthalmol.2015.0789. PMID 25905446
- [Background] Carter SR, Stewart JM, Khan J, Archer KF, Holds JB, Seiff SR, Dailey RA. Infection after blepharoplasty with and without carbon dioxide laser resurfacing. Ophthalmology. 2003 Jul;110(7):1430-2. doi: 10.1016/S0161-6420(03)00447-0. PMID 12867404
- [Background] Saco M, Howe N, Nathoo R, Cherpelis B. Topical antibiotic prophylaxis for prevention of surgical wound infections from dermatologic procedures: a systematic review and meta-analysis. J Dermatolog Treat. 2015 Apr;26(2):151-8. doi: 10.3109/09546634.2014.906547. Epub 2014 Apr 8. PMID 24646178
- [Background] Mangram AJ, Horan TC, Pearson ML, Silver LC, Jarvis WR. Guideline for prevention of surgical site infection, 1999. Hospital Infection Control Practices Advisory Committee. Infect Control Hosp Epidemiol. 1999 Apr;20(4):250-78; quiz 279-80. doi: 10.1086/501620. No abstract available. PMID 10219875
- [Background] Ferneini EM, Halepas S, Aronin SI. Antibiotic Prophylaxis in Blepharoplasty: Review of the Current Literature. J Oral Maxillofac Surg. 2017 Jul;75(7):1477-1481. doi: 10.1016/j.joms.2017.01.025. Epub 2017 Feb 1. PMID 28222277
- [Background] Rogers HD, Desciak EB, Marcus RP, Wang S, MacKay-Wiggan J, Eliezri YD. Prospective study of wound infections in Mohs micrographic surgery using clean surgical technique in the absence of prophylactic antibiotics. J Am Acad Dermatol. 2010 Nov;63(5):842-51. doi: 10.1016/j.jaad.2010.07.029. Epub 2010 Aug 30. PMID 20800320
- [Background] Levender MM, Davis SA, Kwatra SG, Williford PM, Feldman SR. Use of topical antibiotics as prophylaxis in clean dermatologic procedures. J Am Acad Dermatol. 2012 Mar;66(3):445-51. doi: 10.1016/j.jaad.2011.02.005. Epub 2011 Aug 6. PMID 21821310

RESULTS

PARTICIPANT FLOW:
Groups:
- Topical Antibiotic Ointment: The antibiotic arm received either erythromycin or a bacitracin containing ointment, depending on allergies, surgeon preference, and pharmacy availability. Patients were instructed to apply the ointment to the surgical incision(s) 4 times daily for 1 week.
- Topical Non-Antibiotic Ointment: The non-antibiotic ointment arm received mineral oil/petrolatum-based artificial tear ointment with instructions to apply it to the surgical incision(s) 4 times daily for 1 week.
Period: Overall Study
Arm/Group | Topical Antibiotic Ointment | Topical Non-Antibiotic Ointment
Started | 208 | 193
Did Not Proceed With Surgery | 2 | 1
Received Allocated Treatment | 206 | 192
Lost to Follow-up | 5 | 5
Primary Outcome Analyzed | 201 | 187
Completed | 201 | 187
Not Completed | 7 | 6
Not completed — Lost to Follow-up | 5 | 5
Not completed — Did not proceed with surgery | 2 | 1

BASELINE CHARACTERISTICS:
Population: Data not available for 3 participants who did not proceed with surgery.
Groups:
- Total: Total of all reporting groups
Arm/Group | Topical Antibiotic Ointment | Topical Non-Antibiotic Ointment | Total
Number analyzed (Participants) | 206 | 192 | 398
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.5 (16.7) | 63.4 (15.4) | 63.5 (16.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 127 | 112 | 239
  Male | 79 | 80 | 159
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 12 | 29
  Not Hispanic or Latino | 189 | 179 | 368
  Unknown or Not Reported | 0 | 1 | 1
Smoking status [Count of Participants; unit: Participants]
  Yes | 18 | 13 | 31
  No | 188 | 178 | 366
  Unknown | 0 | 1 | 1
High risk for infection [Count of Participants; unit: Participants] — Participants were considered high risk for infection if they had a history of smoking or a medical history of a condition associated with immune suppression, such as diabetes mellitus, infection with human immunodeficiency virus, or autoimmune disease requiring immunosuppressive agents.
  Participants
    Yes | 44 | 47 | 91
    No | 162 | 145 | 307
Asplenia [Count of Participants; unit: Participants]
  Yes | 1 | 0 | 1
  No | 205 | 192 | 397
Autoimmune disease [Count of Participants; unit: Participants]
  Yes | 6 | 2 | 8
  No | 200 | 190 | 390
Diabetes mellitus [Count of Participants; unit: Participants]
  Yes | 24 | 31 | 55
  No | 182 | 161 | 343
Human immunodeficiency virus infection [Count of Participants; unit: Participants]
  Yes | 0 | 4 | 4
  No | 206 | 188 | 394
Malignancy [Count of Participants; unit: Participants]
  Yes | 0 | 2 | 2
  No | 206 | 190 | 396
Organ transplantation [Count of Participants; unit: Participants]
  Yes | 0 | 1 | 1
  No | 206 | 191 | 397
Blepharoplasty [Count of Participants; unit: Participants]
  Yes | 48 | 39 | 87
  No | 158 | 153 | 311
Browplasty [Count of Participants; unit: Participants]
  Yes | 3 | 0 | 3
  No | 203 | 192 | 395
Dacryocystorhinostomy [Count of Participants; unit: Participants]
  Yes | 1 | 6 | 7
  No | 205 | 186 | 391
Ectropion/Entropion repair [Count of Participants; unit: Participants]
  Yes | 25 | 25 | 50
  No | 181 | 167 | 348
Eyelid lesion removal and/or biopsy [Count of Participants; unit: Participants]
  Yes | 36 | 36 | 72
  No | 170 | 156 | 326
Ptosis repair [Count of Participants; unit: Participants]
  Yes | 41 | 43 | 84
  No | 165 | 149 | 314
Reconstruction after Mohs surgery [Count of Participants; unit: Participants]
  Yes | 25 | 22 | 47
  No | 181 | 170 | 351
Orbitotomy [Count of Participants; unit: Participants]
  Yes | 8 | 11 | 19
  No | 198 | 181 | 379
Tarsorrhaphy [Count of Participants; unit: Participants]
  Yes | 3 | 1 | 4
  No | 203 | 191 | 394
Wedge excision [Count of Participants; unit: Participants]
  Yes | 15 | 15 | 30
  No | 191 | 177 | 368

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Surgical Site Infections
Description: The rate of superficial incisional or deep incisional surgical site infection (SSI) of clean and clean-contaminated wounds.
Time Frame: First Post-Operative Visit (~7-14 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Topical Antibiotic Ointment | Topical Non-Antibiotic Ointment
Number analyzed (Participants) | 201 | 187
Participants | 0 | 5
Statistical Analysis 1: Comparison: Topical Antibiotic Ointment vs Topical Non-Antibiotic Ointment; Test type: Superiority; p = 0.025, Fisher Exact; Risk Ratio (RR) = 0.00

2. Secondary Outcome: Number of High Risk Participants With Surgical Site Infections
Description: A secondary outcome is the rate of superficial or deep SSI in participants considered high risk for infection due to comorbidities such as smoking, exogenous immunosuppressive agent use, or medical conditions causing immunosuppression such as diabetes mellitus.
Time Frame: First Post-Operative Visit (~7-14 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Topical Antibiotic Ointment | Topical Non-Antibiotic Ointment
Number analyzed (Participants) | 44 | 47
Participants | 0 | 1

3. Secondary Outcome: Number of Participants With Wound Dehiscence
Description: A secondary outcome recording the rate of wound dehiscence after surgery.
Time Frame: First Post-Operative Visit (~7-14 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Topical Antibiotic Ointment | Topical Non-Antibiotic Ointment
Number analyzed (Participants) | 201 | 187
Participants | 7 | 5
Statistical Analysis 1: Comparison: Topical Antibiotic Ointment vs Topical Non-Antibiotic Ointment; Test type: Superiority; p = 0.77, Fisher Exact; Risk Ratio (RR) = 1.30, 95% CI 2-sided [0.42 to 4.03]

4. Secondary Outcome: Number of Participants With Allergic Contact Dermatitis
Description: A secondary outcome recording the rate of allergic contact dermatitis due to post-operative ointment.
Time Frame: First Post-Operative Visit (~7-14 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Topical Antibiotic Ointment | Topical Non-Antibiotic Ointment
Number analyzed (Participants) | 201 | 187
Participants | 1 | 1
Statistical Analysis 1: Comparison: Topical Antibiotic Ointment vs Topical Non-Antibiotic Ointment; Test type: Superiority; p = 1.00, Fisher Exact; Risk Ratio (RR) = 0.93, 95% CI 2-sided [0.06 to 14.77]

ADVERSE EVENTS:
Time Frame: Adverse events were collected until the final post-operative visit (approximately 3 months).
Description: Among participants who did not proceed with surgery or who had no post-operative follow-up, adverse event data for events specific to the post-operative period (i.e. allergic contact dermatitis or wound dehiscence) were not collected. These participants were excluded from the denominator in determining frequency of these adverse events.
Arm/Group | Topical Antibiotic Ointment | Topical Non-Antibiotic Ointment
All-Cause Mortality (participants affected / at risk) | 0/208 | 0/193
Serious Adverse Events (participants affected / at risk) | 0/208 | 0/193
Other Adverse Events (participants affected / at risk) | 8/208 | 6/193
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Topical Antibiotic Ointment (N=208) | Topical Non-Antibiotic Ointment (N=193)
Allergic contact dermatitis (Skin and subcutaneous tissue disorders) | 1/201 (1) | 1/187 (1) — Allergic contact dermatitis at the surgical site.
Wound dehiscence (Skin and subcutaneous tissue disorders) | 7/201 (7) | 5/187 (5) — Dehiscence of the surgical wound.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2018-09-09): https://cdn.clinicaltrials.gov/large-docs/11/NCT03199911/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-01): https://cdn.clinicaltrials.gov/large-docs/11/NCT03199911/SAP_001.pdf